CLINICAL TRIAL: NCT06625450
Title: TOFACITINIB COMPARED TO TOFACITINIB WITH MESALAMINE FOR MAINTENANCE OF REMISSION IN ULCERATIVE COLITIS: A RANDOMIZED CONTROLLED TRIAL
Brief Title: TOFACITINIB vs TOFACITINIB WITH MESALAMINE IN ULCERATIVE COLITIS
Status: Not yet recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: Post Graduate Institute of Medical Education and Research, Chandigarh (Other)
Responsible Party: Principal Investigator, Beenal Dhooria, Senior Resident (DM Fellow), Post Graduate Institute of Medical Education and Research, Chandigarh
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: TOME
Record Dates: First submitted 2024-10-02; First posted 2024-10-03 (Actual); Last update posted 2024-10-03 (Actual); Status verified 2024-10

CONDITIONS: Ulcerative Colitis
MeSH Terms: conditions — Colitis, Ulcerative | interventions — tofacitinib; Mesalamine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Tofacitinib (Active Comparator): Mesalamine will be withdrawn while tofacitinib will be continued during maintenance of remission of the disease
  Interventions: Drug: Tofacitinib
- Tofacitinib plus mesalamine (Active Comparator): Both mesalamine and tofacitinib will be continued during maintenance of remission of the disease
  Interventions: Drug: Tofacitinib plus mesalamine

INTERVENTIONS:
Drug: Tofacitinib — Tofacitinib alone will be continued at a dose of 11 mg once a day
  Arms: Tofacitinib
Drug: Tofacitinib plus mesalamine — Both tofacitinib 11 mg once a day and mesalamine will be continued
  Arms: Tofacitinib plus mesalamine

SUMMARY:
All the trials using tofacitinib for maintenance of remission in UC have allowed the use of concomitant therapies except glucocorticoids. Mesalamine, a drug used in mild-to-moderate UC is often continued in patients receiving other drugs for maintenance. In this study, we plan to compare the effect of withdrawing mesalamine and continuing monotherapy with tofacitinib versus continuing dual therapy with tofacitinib and mesalamine. We hypothesize that the continuation of tofacitinib monotherapy after withdrawing mesalamine will be as efficacious and safe as continuation of the combination in remission maintenance in UC.

DETAILED DESCRIPTION:
Inflammatory bowel disease (IBD) is a chronic inflammatory condition of bowel having a relapsing and remitting course. It has two major forms: ulcerative colitis (UC) and Crohn's disease (CD). Other less common forms include microcytic colitis, primary collagenous colitis and lymphocytic colitis. Ulcerative colitis is a form of IBD in which there is continuous involvement of the colon with the inflammation initiating from the rectum and then progressively involving variable lengths of the large intestine. Both genetic predisposition and environmental factors play a role. A dysregulated immune response, gut microbiota and epithelial barrier defects are implicated in the pathogenesis of UC.

The usual presentation is bloody diarrhoea. Diagnosis is based on clinical, endoscopic and histological findings. The aim of treatment in ulcerative colitis is to induce clinical, biochemical and endoscopic remission and to maintain it on a long-term. Various treatment options include 5-ASA, glucocorticoids, thiopurines, biologicals and small molecules. 5-ASA is used both in inducing and maintaining remission in UC. As per the American Gastroenterology Association (AGA) guidelines, 5-ASA is used as the first line agent for inducing remission in mild to moderate UC (1). It has also been extensively evaluated in the maintenance of remission (2). In an initial multicentre study, 264 subjects with UC in remission for 1 month were randomized into a mesalamine and a placebo arm. Endoscopic remission at 6 months was the primary endpoint defining treatment success. In both the intention-to-treat and per protocol analyses, mesalamine was significantly better than placebo for remission maintenance the end of 6 months. Since then, several studies have demonstrated the efficacy of different preparations of mesalamine in maintaining remission in ulcerative colitis.

Tofacitinib has also been studied in the OCTAVE trials for both induction and maintenance of remission in UC. In the OCTAVE induction 1 and 2 trials, tofacitinib was compared to placebo for induction of remission in moderate-to-severe UC and it was found to be better than placebo. Various meta-analyses also confirmed the same. The OCTAVE sustain proved tofacitinib to be better than placebo in maintaining UC in remission at both the studied doses (10 mg twice daily and 5 mg twice daily). All the trials using tofacitinib for maintenance of remission in UC have allowed the use of concomitant therapies except glucocorticoids. Mesalamine, a drug used in mild-to-moderate UC is often continued in patients receiving other drugs for maintenance. Recent guidelines have emphasised the importance of low-cost healthcare as there is increasing pressure on healthcare budgets worldwide (3). A study in the United Kingdom suggested that mesalamine accounts for up to 25% of the total healthcare costs in UC, with an average annual maintenance prescription estimated to be £740 or €850 (4). While mesalamine is safe and well-tolerated, it has rare but serious idiosyncratic adverse effects including pancreatitis. Around 3% of patients even report a paradoxical worsening of diarrhoea (5). The negative impact of polypharmacy must also be taken into consideration, with non-compliance often linked to higher pill burdens (6). In fact, the burden of a more complex medication regimen has been associated with poorer outcomes in both UC with real-world compliance as low as 50% (7). Furthermore, compliance to topical 5-ASA therapy is even worse than oral therapy (8). Thus, there is a clear need to explore the withdrawal of 5-ASA from the UC treatment regimen.

Two studies have evaluated the outcomes of withdrawal of oral 5-ASA in patients concomitantly treated with immunomodulators. Both studies showed no difference in relapse rates between patients with ulcerative colitis receiving either azathioprine monotherapy or combination of azathioprine and oral 5-ASA therapy with better compliance in azathioprine monotherapy group (9, 10). No randomized controlled trial (RCT) has yet evaluated the withdrawal of 5-ASA in patients treated with either biologic therapy or tofacitinib. However, a recent cohort study from two national population-based databases (from the United States and Denmark) showed no increase in the risk of adverse clinical events after withdrawing oral 5-ASA within 90 days of initiating anti-TNF therapy compared to those who continued 5-ASA (11). No RCT or prospective study has evaluated the outcome of 5-ASA withdrawal in patients receiving tofacitinib therapy. Indirect evidence from subgroup analysis of RCTs suggests that concomitant 5-ASA therapy does not increase the likelihood of maintaining clinical remission after escalation to tofacitinib (12).

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed cases of UC by endoscopy and biopsy
* Patients in clinical remission for at least 3 months on Tofacitinib and mesalamine

Exclusion Criteria:

* Incomplete evaluation
* Uncertain diagnosis
* Active disease
* Subjects with Crohn's disease, microscopic colitis and collegenous colitis or IBD-U
* Unwilling to participate in study
* Pregnant and lactating women or those who are planning pregnancy in the forthcoming 2 years
* Patients with any suspected or proven malignancy
* Subjects with severe comorbidities
* Prior history of venous thromboembolism.
* Subjects undergoing major surgery
* Myocardial infarction within previous 3 months
* Heart failure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 75 (Estimated)
Dates: Start 2024-10 (Estimated); Primary Completion 2025-12 (Estimated); Study Completion 2026-01 (Estimated)

PRIMARY OUTCOMES:
Time to relapse of colitis | 12 months
  Relapse of ulcerative colitis will be diagnosed based on the study subject's clinical findings

SECONDARY OUTCOMES:
Serum biomarker C-reactive protein | 12 months
  Changes in the level of serum biomarker C-reactive protein
Serum biomarker calprotectin | 12 months
  Changes in the level of serum biomarker calprotectin
Physician global assessment | 12 months
  The physician will assess the overall clinical condition of the subject on a visual analog scale from 0 to 100
Adverse effects | 12 months
  The adverse effects of the study drugs (venous thromboembolism, nasopharyngitis, diarrhea) and any other patient-reported adverse effects

IPD SHARING:
Plan to Share IPD: Yes
Anonymized data will be shared after publication on reasonable request.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: After publication...for 2 years